CLINICAL TRIAL: NCT04349007
Title: Integrating the Power of Peanuts Into School Feeding Programs in Ghana
Brief Title: Power of Peanuts School Feeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Ghana (Other); Project Peanut Butter, Ghana (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202011110
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: School Feeding Programs; Nutrition Supplements
MeSH Terms: interventions — Milk

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single (Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard meal (Active Comparator): local porridge with a vitamin and mineral sprinkle powder that will be mixed in
  Interventions: Dietary Supplement: Standard meal
- School food ready-to-use (Experimental): peanut-based school food ready-to-use
  Interventions: Dietary Supplement: School food ready-to-use
- School food ready-to-use plus Milk (Experimental): peanut-based school food ready-to-use with milk
  Interventions: Dietary Supplement: School food ready-to-use plus Milk

INTERVENTIONS:
Dietary Supplement: Standard meal — local porridge with a vitamin and mineral sprinkle powder that will be mixed in after cooking
  Arms: Standard meal
Dietary Supplement: School food ready-to-use — 80 gram per day sachet containing peanut paste with oil, sugar, cowpea, maize, and vitamin and minerals
  Arms: School food ready-to-use
Dietary Supplement: School food ready-to-use plus Milk — 80 gram per day sachet containing peanut paste with oil, sugar, cowpea, non-fat dried milk and vitamin and minerals
  Arms: School food ready-to-use plus Milk

SUMMARY:
This will be a two-phase protocol. Phase 1 will include the development of the peanut-based school food, and a small formative research study on the acceptability and consumption of the school food study intervention. This will occur among children 5-12 yr in the Mion district, 60 school aged children between 6-12 years old will be recruited to participate in a 3 week consumption and acceptability study. An integral part of the food development process is acceptability testing. A child must like and want to eat a new food if it is to be consumed as prescribed and effective in potential improving linear growth and cognitive performance. This study will confirm that food developed for the school feeding clinical trial will be consumed as dosed and what additional snack food offerings may be useful in encouraging consumption.

Phase 2 will be a individually randomized, investigator blinded, controlled clinical effectiveness trial of a peanut-based school meal with and without milk powder compared to a control meal for linear growth and cognitive performance. 880 children 5 to 12 years old, healthy, enrolled in primary school, including kindergarten at 6 selected schools in the Mion district will be randomized to receive one of three school foods, a peanut-based food with milk, a peanut-based food without milk and a control group composed of commonly available tuber/cereal. The sample size accounts for up to 15% attrition for a final sample size of 750 with a total 250 eligible children enrolled in each group. Enrolled children will receive the meal daily during the school lunch period for an entire school year. At enrollment and upon completion, anthropometric measurements and body composition data will be collected and a tablet- based, language independent cognitive test battery will be administered. Basic demographic information and school attendance information will be collected as well.

ELIGIBILITY:
Inclusion Criteria:

* Healthy school children

Exclusion Criteria:

* severe malnutrition
* chronic debilitation disease
* peanut or milk allergy
* not attending school

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 880 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Fluid cognition as measured by tests in NIH toolbox | 10 months
  Dimensional change card Sort, performance score
Fluid cognition as measured by tests in NIH toolbox | 10 months
  Flanker inhibitory control and attention, performance score
Fluid cognition as measured by tests in NIH toolbox | 10 months
  List sorting working memory, performance score
Fluid cognition as measured by tests in NIH toolbox | 10 months
  Pattern comparison processing speed, performance score

SECONDARY OUTCOMES:
Height-for-age Z | 10 months
  difference between enrollment and end of study height-for-age z score
Change in body mass index | 10 months
  difference between enrollment and end of study body mass index

CONTACTS AND LOCATIONS:
Overall Officials: Mark Manary, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Project Peanut Butter, Tamale, Ghana

REFERENCES:
- [Derived] Stephenson KB, Wegner DR, Hershey TG, Doty T, Davis E, Steiner-Asiedu M, Saalia FK, Shani I, Manary MJ. Effect of Peanut Paste-based Ready-to-use School Meals With and Without Milk on Fluid Cognition in Northern Ghana: A Randomized Controlled Trial. Am J Clin Nutr. 2023 Oct;118(4):782-791. doi: 10.1016/j.ajcnut.2023.08.001. Epub 2023 Aug 9. PMID 37567391